CLINICAL TRIAL: NCT06735404
Title: Regular and Unplanned Care Adaptive Dashboard for Cross-border Emergencies (RAPIDE): The Feasibility of a Hybrid Care Model
Brief Title: RAPIDE: The Feasibility of a Hybrid Care Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-17762
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Type 2; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hybrid care (Experimental)
  Interventions: Other: Hybrid care

INTERVENTIONS:
Other: Hybrid care — The hybrid care model will consist of a combination of digital tools and/or task shifting of certain healthcare providers. Examples are:
  * Telemonitoring: patients perform self-measurements through e.g. sensors, wearables, or (mobile) applications to get insight in their health status (supporting self-management) and report this to their healthcare provider(s), when relevant
  * Teleconsultation: patients communicate with their healthcare provider(s) remotely
  * Personal health portals and self-management applications
  * Online prescription requests: patients request prescription online

SUMMARY:
Rationale: During cross-border health emergencies, such as seen with the COVID-19 pandemic, health and care services are rapidly being overwhelmed by high numbers of patients requiring care, leading to stretches in the whole healthcare system. Delays and backlogs in regular care, as the result of the stretched health care services, leave millions of patients with regular care needs unattended, resulting in disastrous healthcare outcomes. If disastrous healthcare outcomes across the population are to be avoided, healthcare systems must become more robust, resilient, and flexible in the face of future health emergencies and allow for rapid changes in the care delivery services.

Objective: To evaluate the feasibility of delivering a hybrid care model alongside care as usual through observations, and questionnaires and interviews on patient reported views, opinions, and experiences. This hybrid care model aims to reduce the burden on health and care systems during a health emergency, decrease the need to scale down regular care, and ensure patient safety and quality of care.

Study design: One year cohort study, using observations, questionnaires, and interviews.

Study population: Patients with type 2 diabetes and/or chronic heart failure with comorbidities and/or having a high care consumption according to the treating general practitioner.

Intervention: The hybrid care model will consist of a combination of digital tools and/or task shifting of certain healthcare providers. Examples are:

* Telemonitoring: patients perform self-measurements through e.g. sensors, wearables, or (mobile) applications to get insight in their health status (supporting self-management) and report this to their healthcare provider(s), when relevant
* Teleconsultation: patients communicate with their healthcare provider(s) remotely
* Personal health portals and self-management applications
* Online prescription requests: patients request prescription online Main study parameters/endpoints: The impact of the hybrid care model on patient reported experiences (PREMs) and patient reported outcomes (PROMs).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Evaluating the feasibility of this hybrid care model will only be done through observations, questionnaires, and interviews at home (during three home visits at baseline, after six months, and after one year). No invasive (physical) procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

Patients with type 2 diabetes mellitus, WITH:

* At least 2 different types of chronic comorbidities (as defined in the list of chronic comorbidities); AND
* A high number of medical consultations at the GP practice and/or referrals to the hospital in the last 24 months, as identified by the clinical expertise of the treating GP.

Patients with chronic heart failure, WITH:

* At least 2 different types of chronic comorbidities (as defined in the list of chronic comorbidities); AND
* A high number of medical consultations at the GP practice and/or referrals to the hospital in the last 24 months, as identified by the clinical expertise of the treating GP.

Exclusion Criteria:

* Terminally ill patients
* Comorbidity of a severe psychiatric disorder (i.e. psychosis-related disorders, dementia, and bipolar disorder)
* Patients who are cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The impact of the hybrid care model on patient reported experiences (PREMs) and patient reported outcomes (PROMs), using the PaRIS questionnaire. | At enrolment, at six months after enrolment, and at twelve months after enrolment.

SECONDARY OUTCOMES:
Episodes of care consumption, using patient chart reviews | At baseline and 12 months after enrolment

OTHER OUTCOMES:
Acceptability and feasibility from the perspective of patients, informal caregivers, and healthcare professionals, using observations and interviews | Six and twelve months after enrolment.
  Through observations and interviews, the investigators will evaluate the extent to which the hybrid care model is acceptable and feasible for patients, informal care givers, and healthcare professionals.
Implementation feasibility, using observations and interviews | Six and twelve months after enrolment.
  Through observations and interviews, the investigators will evaluate the extent to which the new hybrid care model is practically feasible to implement (facilitators and barriers of implementation).
Changes in practice organisation and care delivery, using observations and interviews | Six and twelve months after enrolment.
  Through observations and interviews, the investigators will evaluate the extent to which the new hybrid care model initiates changes in practice organisation and care delivery.

CONTACTS AND LOCATIONS:
Locations (4):
- Accademia Italiana Cure Primarie, Verona, Italy
- University of Malta, Valletta, Malta
- Radboud University Medical Center, Nijmegen, Netherlands
- Community Health Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No